CLINICAL TRIAL: NCT01239056
Title: Prospective Evaluation of the Clinical Utility of Pseudocyst Drainage With Metal Stent
Brief Title: Evaluation of Pancreatic Pseudocyst Drainage With a Metal Stent
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: Pancreatic Pseudocyst
Record Dates: First submitted 2010-11-05; First posted 2010-11-11 (Estimated); Results first posted 2015-08-21 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-08

CONDITIONS: Pancreatic Pseudocysts
MeSH Terms: conditions — Pancreatic Pseudocyst | interventions — Endoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pancreatic Pseudocysts: All adult patients who have a clinical indication to undergo an endoscopic drainage of a pancreatic pseudocyst.
  Interventions: Procedure: Endoscopy

INTERVENTIONS:
Procedure: Endoscopy — Endoscopic drainage of a pancreatic pseudocyst using a metal stent per medical indication.

SUMMARY:
The purpose of this study is to study the evaluation of the effectiveness of endoscopic Pancreatic Pseudocyst drainage using a metal stent.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 years or older
2. Subject has pancreatic pseudocyst
3. Subject has medical indication for drainage of the pancreatic pseudocyst
4. Subject must be able to give informed consent

Exclusion Criteria:

1. Any contraindication to endoscopic pseudocyst drainage
2. Subject is unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have a medical indication for endoscopic drainage of pancreatic pseudocyst and are referred for the procedure as part of their standard medical care will be considered for the study.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2009-08; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter V draganov, MD, Principal Investigator — University of Florida
Locations (1):
- Shands UF Endoscopy, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 22 signed informed consents, however after Endoscopic ultrasound imaging, 2 participants were excluded due to characteristics of the cyst cavity. Therefore, 20 participants underwent transgastric drainage of pancreatic pseudocysts by use of the fully covered self-expanding metal stents (CSEMS).
Groups:
- Pancreatic Pseudocysts: Patients underwent Endoscopic Ultrasound-guided pseudocyst transmural drainage using fully covered self-expanding metal stents (CSEMS). Next, patients underwent an Endoscopic retrograde cholangiopancreatography to evaluate for Pancreatic duct (PD) disruption. Patients then received an abdominal CT to assess pancreatic pseudocyst resolution. If complete resolution was noted, all stents were subsequently removed. If the pseudocyst was not resolved, stent removal was deferred and follow-up CTs were obtained at 2 to 4 week intervals until radiographic resolution was achieved.
Period: Overall Study
Arm/Group | Pancreatic Pseudocysts
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pancreatic Pseudocysts
Number analyzed (Participants) | 20
Age, Continuous [Mean (Full Range); unit: years] | 57 [34 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 15
Pseudocyst diameter [Mean (Full Range); unit: centimeters] | 13.4 [5.5 to 23]

OUTCOME MEASURES:

1. Secondary Outcome: Resolution of Pancreatic Pseudocyst After Placement of Fully Covered Self-expanding Metal Stent (CSEMS).
Time Frame: 6 to 12 weeks after baseline
Measure: Number; unit: participants
Groups:
- Pancreatic Pseudocysts: Patients underwent Endoscopic Ultrasound-guided pseudocyst transmural drainage using fully covered self-expanding metal stents (CSEMS). Next, patients underwent Endoscopic retrograde cholangiopancreatography to evaluate for Pancreatic duct (PD) disruption. Patients then received an abdominal CT to assess pancreatic pseudocyst resolution. If complete resolution was noted, all stents were subsequently removed. If the pseudocyst was not resolved, stent removal was deferred and follow-up CTs were obtained at 2 to 4 week intervals until radiographic resolution was achieved.
Arm/Group | Pancreatic Pseudocysts
Number analyzed (Participants) | 20
participants
  Resolution of Pseudocyst | 17
  Unresolved Pseudocyst | 3

2. Primary Outcome: Technical Success of Endoscopic Ultrasound-guided Single-access Pseudocyst Drainage With a Fully Covered Self-expanding Metal Stent ; Anchored With a Double Pigtail Plastic Stent Inserted Through the Metal Stent Lumen
Description: Technical success was evaluated by the ability to achieved pseudocyst drainage after endoscopically placing a Fully Covered Self-expanding Metal Stent in the pseudocyst .
  Technical failure was evaluated by the inability to fully drain the pancreas pseudocyst after endoscopically placing a Fully Covered Self-expanding Mental Stent in the pseudocyst.
Time Frame: baseline
Measure: Number; unit: participants
Arm/Group | Pancreatic Pseudocysts
Number analyzed (Participants) | 20
participants
  technical success | 20
  technical failure | 0

3. Secondary Outcome: Adverse Events
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Pancreatic Pseudocysts
Number analyzed (Participants) | 20
participants
  Pseudocyst infection requiring surgery | 2
  Posttransmural drainage fever | 1
  PostEndoscopic retrograde cholangiopancreatography | 1

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Pancreatic Pseudocysts
Serious Adverse Events (participants affected / at risk) | 2/20
Other Adverse Events (participants affected / at risk) | 1/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pancreatic Pseudocysts (N=20)
pseudocyst infection requiring surgery (Gastrointestinal disorders) | 2 (2) — Major complication from transmural drainage
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pancreatic Pseudocysts (N=20)
posttransmural drainage fever (Gastrointestinal disorders) | 1 (1)
post-ERCP pancreatitis (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes